CLINICAL TRIAL: NCT05285085
Title: Real World Evidence Study for Assessing Statin Use for Primary and Secondary Prevention of Cardiovascular Disease in Primary Care in Brazil
Brief Title: Real World Evidence Study of Statin Use in Brazil
Acronym: RWE-Statins
Status: Completed | Type: Observational
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: epHealth (Unknown); Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: 53194121.0.0000.0071
Record Dates: First submitted 2022-03-02; First posted 2022-03-17 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2022-03

CONDITIONS: Cardiovascular Diseases; Myocardial Infarction; Stroke; Hypertension; Diabetes Mellitus; Dyslipidemias
Keywords: cardiovascular diseases; primary prevention; secondary prevention; statins
MeSH Terms: conditions — Cardiovascular Diseases; Myocardial Infarction; Stroke; Hypertension; Diabetes Mellitus; Dyslipidemias | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors; Simvastatin; Rosuvastatin Calcium; Atorvastatin; pitavastatin; Pravastatin; Lovastatin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Secondary prevention: Individuals with previous myocardial infarction and/or stroke
  Interventions: Drug: Statin
- Primary prevention: Individuals with hypertension, diabetes and/or dyslipidemia
  Interventions: Drug: Statin
- Unknown diagnosis: Individuals without a previous myocardial infarction and/or stroke or a diagnosis of hypertension, diabetes and/or dyslipidemia
  Interventions: Drug: Statin

INTERVENTIONS:
Drug: Statin — Statin use
  Other Names: simvastatin; calcium rosuvastatin; atorvastatin; pitavastatin; pravastatin; lovastatin; rosuvastatin

SUMMARY:
A cross-sectional real-world data study designed to assess the use of statins in individuals assisted within the primary care system in Brazil.

DETAILED DESCRIPTION:
Considering the high cardiovascular risk associated to high cholesterol levels, assessing the use of statins in secondary prevention as well as primary prevention individuals in real world settings is key to enable public health policy improvements.

The aim of the present study is to assess statins use in primary and secondary prevention individuals assisted by community care workers in the primary care system in Brazil, using a free real world data collection tool (epHealth database). Evaluating factors associated with statins use as well as high dose statins use are also objectives of the study.

ELIGIBILITY:
Inclusion Criteria:

* All individuals aged 18 years or older registered on the epHealth database

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All individuals aged 18 years or older registered on the epHealth database will be used in this study.
Sampling Method: Non-Probability Sample
Enrollment: 2133900 (Actual)
Dates: Start 2021-11-19 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Statin use on secondary prevention | Baseline
  Proportion of patients with previous myocardial infarction and/or stroke on statin use
Statin use on primary prevention | Baseline
  Proportion of patients with hypertension, diabetes and/or dyslipidemia on statin use

SECONDARY OUTCOMES:
Statin use on patients with previous myocardial infarction | Baseline
  Proportion of patients with previous myocardial infarction on statin use
Statin use on patients with previous stroke | Baseline
  Proportion of patients with previous stroke on statin use
High dose statin use on secondary prevention | Baseline
  Proportion of patients with previous myocardial infarction and/or stroke on high dose statin use
High dose statin use on patients with previous myocardial infarction | Baseline
  Proportion of patients with previous myocardial infarction on high dose statin
High dose statin use on patients with stroke | Baseline
  Proportion of patients with previous stroke on high dose statin
Statin use on patients with diabetes | Baseline
  Proportion of patients with diabetes on statin use
Statin use on patients with hypertension | Baseline
  Proportion of patients with hypertension on statin use
Statin use on patients with dyslipidemia | Baseline
  Proportion of patients with dyslipidemia on statin use
High dose statin use on patients with diabetes | Baseline
  Proportion of patients with diabetes on high dose statin
High dose statin use on patients with hypertension | Baseline
  Proportion of patients with hypertension on high dose statin
High dose statin use on patients with dyslipidemia | Baseline
  Proportion of patients with dyslipidemia on high dose statin
Statin use on patients with unknown diagnosis | Baseline
  Proportion of patients without previous myocardial infarction and/or stroke or a diagnosis of hypertension, diabetes and/or dyslipidemia on statin use
High dose statin use on patients with unknown diagnosis | Baseline
  Proportion of patients without previous myocardial infarction and/or stroke or a diagnosis of hypertension, diabetes and/or dyslipidemia on high dose statin use

CONTACTS AND LOCATIONS:
Overall Officials: M. Julia Machline-Carrion, PhD, Principal Investigator — epHealth
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
No plan

REFERENCES:
- [Result] Machline-Carrion MJ, Girotto AN, Nieri J, Pereira PM, Monfardini F, Forestiero F, Raupp P, Roveda F, Santo K, Berwanger O, Santos RD. Assessing statins use in a real-world primary care digital strategy: a cross-sectional analysis of a population-wide digital health approach. Lancet Reg Health Am. 2023 Jun 22;23:100534. doi: 10.1016/j.lana.2023.100534. eCollection 2023 Jul. PMID 37497398
- [Result] Santo K, Santos RD, Girotto AN, Nieri J, Monfardini F, Raupp P, Pereira PM, Berwanger O, Machline-Carrion MJ. Statins use for primary prevention of cardiovascular disease: A population-based digitally enabled real-world evidence cross-sectional study in primary care in Brazil. J Clin Lipidol. 2024 May-Jun;18(3):e384-e393. doi: 10.1016/j.jacl.2024.02.005. Epub 2024 Feb 20. PMID 38431498